CLINICAL TRIAL: NCT00731965
Title: Multicenter Randomized Clinical Trial in Patients With Juvenile Idiopathic Arthritis: Safety and Efficacy of Vaccination With Live Attenuated Measles, Mumps, Rubella Vaccine
Brief Title: Safety and Efficacy of Measles, Mumps, Rubella Vaccination in Juvenile Idiopathic Arthritis
Acronym: VAART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: N.M. Wulffraat (Other)
Collaborators: University Medical Center Groningen (Other); Amsterdam UMC, location VUmc (Other); Maastricht University Medical Center (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor-Investigator, N.M. Wulffraat, associate professor, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: VAART; ISRCTN12271664
Record Dates: First submitted 2008-08-06; First posted 2008-08-11 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: Arthritis, Juvenile Rheumatoid; Measles-Mumps-Rubella Vaccine; Serology; Lymphocytes
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Measles, mumps, rubella booster vaccination within 3 months after randomisation
  Interventions: Biological: Measles, Mumps, Rubella vaccination
- 2 (No Intervention): Booster vaccination performed by regular health authorities at age 9; at least 1 year after randomisation

INTERVENTIONS:
Biological: Measles, Mumps, Rubella vaccination — Dosage: 1 dose MMR vaccine, containing 5000 p.f.u. (plaque forming unit) life attenuated mumps virus (Jeryl-Lynn-strain), 1000 p.f.u. life attenuated measles virus (Moraten-strain) and 1000 p.f.u. life attenuated rubella virus (Wistar RA 27/3-strain) + 0.5 ml solution fluid Dosage form: subcutaneously frequency: once
  Other Names: RVG 17654, BMR-NVI
  Arms: 1

SUMMARY:
Background:

The safety of vaccination in patients with autoimmune diseases using immune suppressive therapy is often discussed. Previous studies in Juvenile Idiopathic Arthritis (JIA) patients showed no increase in disease activity after immunisation with dead vaccines. The safety of the live attenuated Measles, Mumps, Rubella (MMR) vaccination was assessed retrospectively in JIA patients and no increase in disease activity was found. However, this must be prospectively confirmed. In addition, it is unknown whether vaccination is effective, since the immune response to vaccination may be diminished due to immunosuppressive therapy for the underlying disease. Finally, the influence of MMR vaccination on the immune system of JIA patients has not been studied. Among others, regulatory T-cells (Tregs) should control the immune response and prevent destructive autoimmune responses after environmental triggers such as vaccination.

Objective:

The aim of the present study is to investigate the safety and efficacy of the MMR booster vaccination and its influence on immune regulatory mechanisms in children with Juvenile Idiopathic Arthritis.

Method:

JIA patients aged 4 to 8 years and treated by the pediatric rheumatology units from various University Medical Centers in the Netherlands, are asked to participate in a prospective study. In the Netherlands, measles-mumps-rubella (MMR) vaccination is included in the National Vaccination Program and is normally administered at age 9. Included patients will be randomised for early vaccination (age group 4 to 8yr at entry of the study) or at age 9 as is routinely done according to the National Vaccination Program. Prior to and after vaccination the investigators will assess disease activity and collect blood.

Outcome:

During a 12 month follow-up period the investigators will register disease activity and side-effects at different moments in time to determine safety of vaccination. The efficacy of the vaccine will be studied according to antibody levels and function against measles, mumps and rubella in the blood. Tregs will be isolated and their functionality will be determined using the blood cells collected during follow-up. This enables us to study the role influence of vaccination on regulatory mechanisms in our immune system.

ELIGIBILITY:
Inclusion Criteria:

* all subtypes of JIA according to ILAR criteria
* ages 4 to 9 (before the scheduled booster, normally administered at age 9 in the Netherlands)
* 5 healthy adults (aged 18 to 65y)

Exclusion Criteria:

* use of Infliximab (Remicade, anti-Tumor Necrosis Factor (TNF) alpha therapy).
* primary immunodeficiency
* fever less than 48 hour prior to vaccination (vaccination will be postponed for 1 month)
* evidence of viral or bacterial infection less than 48hours prior to vaccination (vaccination will be postponed for 1 month)
* methylprednisolone pulse therapy less than 1 month prior to vaccination (vaccination will be postponed for 1 month)
* transfusion of blood or blood products (e.g. intravenous immunoglobulins (IVIG)) in the 3 months prior to vaccination (vaccination will be postponed for 3 months)

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
JIA disease activity, defined by the core set criteria for JIA and number of flares | baseline and after 3, 6,9,12 months

SECONDARY OUTCOMES:
Immunological reaction to MMR vaccination and regulatory mechanisms induced by MMR, measured by number and function of MMR-specific T cells and cytokine profiles | baseline, 3 and 12 months
  immunogenicity measuring antibody titers and T cell profileration to rubella virus

CONTACTS AND LOCATIONS:
Overall Officials: Nico M. Wulffraat, MD;PhD, Principal Investigator — UMC Utrecht
Locations (5):
- Netherlands (5):
  - Academic hospital Maastricht, Maastricht, Limburg
  - University Medical Center Groningen, Beatrix Children's Hospital, Groningen, Provincie Groningen
  - University Medical Center Utrecht, Wilhelmina Children's Hospital, Utrecht, Utrecht
  - VU University Medical Center Amsterdam, Amsterdam
  - Erasmus Medical Center Rotterdam; sophia Children's Hospital, Rotterdam

REFERENCES:
- [Background] Heijstek MW, Pileggi GC, Zonneveld-Huijssoon E, Armbrust W, Hoppenreijs EP, Uiterwaal CS, Kuis W, Wulffraat NM. Safety of measles, mumps and rubella vaccination in juvenile idiopathic arthritis. Ann Rheum Dis. 2007 Oct;66(10):1384-7. doi: 10.1136/ard.2006.063586. Epub 2007 Feb 6. PMID 17284544
- [Background] Zonneveld-Huijssoon E, Ronaghy A, Van Rossum MA, Rijkers GT, van der Klis FR, Sanders EA, Vermeer-De Bondt PE, Hoes AW, van der Net JJ, Engels C, Kuis W, Prakken BJ, Van Tol MJ, Wulffraat NM. Safety and efficacy of meningococcal c vaccination in juvenile idiopathic arthritis. Arthritis Rheum. 2007 Feb;56(2):639-46. doi: 10.1002/art.22399. PMID 17265499
- [Result] Heijstek MW, Kamphuis S, Armbrust W, Swart J, Gorter S, de Vries LD, Smits GP, van Gageldonk PG, Berbers GA, Wulffraat NM. Effects of the live attenuated measles-mumps-rubella booster vaccination on disease activity in patients with juvenile idiopathic arthritis: a randomized trial. JAMA. 2013 Jun 19;309(23):2449-56. doi: 10.1001/jama.2013.6768. PMID 23780457